CLINICAL TRIAL: NCT03935828
Title: Effect of Topical Sinonasal Antibiotics in Post-Surgical Patients With an Acute Exacerbation of Chronic Rhinosinusitis
Brief Title: Effect of Topical Sinonasal Antibiotics
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI and Record Owner are no longer at our institution
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2018.0060.
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); Antibiotic Side Effect
Keywords: chronic rhinosinusitis; topical sinonasal antibiotics; randomized controlled trial
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Randomized to oral versus topical antibiotics
Who Masked: Outcomes Assessor
Masking Description: Endoscopic sinus scores will be graded by blinded assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Sinonasal Antibiotics (Experimental): For topical antibiotics, the compounding pharmacy will use pre-determined doses using data extrapolated from oral and intravenous doses and data that has detailed the effect of the medication on solubility, pH, and particle properties. Provider choice of topical antibiotics includes Mupirocin 0.4mg/ml, Vancomycin 1mg/ml, Tobramycin 0.7mg/ml, Levofloxacin 0.4mg/ml, and Amphotericin B 20mcg/ml, all to be prescribed for 21 days, applied twice a day. Although the dosing schedule for these topical antibiotics has not been definitively studied, the majority of the data supports a range from two to three times daily for three to four weeks. Patients will be instructed by the pharmacist how to dissolve the cream, powder, or vial of antibiotic in saline, and to irrigate each nostril with 120 ml total. Doses will not be varied during the study period.
  Interventions: Drug: Oral versus topical antibioitics
- Oral Antibiotics (Active Comparator): Oral antibiotics will be prescribed for 21 days, as available (albeit limited) evidence recommends antimicrobial therapy in CRS for at least 3 weeks. For oral antibiotics, the choices providers will be given include: Augmentin 500 mg every 12 hours, Cefuroxime 500 mg every 12 hours, Clarithromycin 500 mg every 6 hours, Levofloxacin 500 mg once daily, or Clindamycin 300 mg every 6 hours, as these are standard of care for treatment of Chronic Rhinosinusitis.
  Interventions: Drug: Oral versus topical antibioitics

INTERVENTIONS:
Drug: Oral versus topical antibioitics — Previously described in two arms

SUMMARY:
In this study, patients who have had previous endoscopic sinus surgery and present with an acute exacerbation of chronic rhinosinusitis will be offered endoscopic-guided, culture-directed antibiotic therapy. They will then be randomized to receive oral or intranasal topical antibiotics. Both of these are considered standard of care, but there is some limited data suggesting superiority of topical antibiotics especially if guided by culture and in patients who have undergone previous surgery. However, a study that directly compares the two has not been published. Modified Lund-Kennedy endoscopic finding scores and subjective SNOT-22 questionnaires will be collected before and at 3-4 weeks after treatment. Medication-related sided effects will be noted and analyzed. After 6-8 month follow-up, we will analyze the rate of recurrence of exacerbations, need for further antibiotics, need for revision surgery, and SNOT-22 scores based on oral versus topical antibiotic treatment. Our objective is to evaluate both short and long-term response to both oral and topical administration of antibiotics in this patient population in order to determine if either route of administration is superior to the other.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have documented CRS refractory to initial medical management and have undergone sinus surgery (opening of at least one sinus ostium, exclusive of sole balloon dilation), and those with an acute exacerbation of CRS with sinus mucopurulence on exam.

Exclusion Criteria:

* Patients less than 18 years of age, and those that have taken an antibiotic regimen in the previous 2 weeks before culture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
SNOT-22 | Baseline, 3-4 weeks after initiation, and at 6-8 months
  Patient-centered, validated 22-item questionnaire assessing SinoNasal outcomes

SECONDARY OUTCOMES:
Modified Lund-Kennedy Score | Baseline and 3-4 weeks after initiation
  Endoscopic grading score of sinonasal inflammation
Antibiotic Side Effect Questions | 3-4 weeks after initiation
  Asking about adverse side effects
Final Questions | 6-8 months
  Asking about recurrence of infections, further need for antibiotics and surgeries

IPD SHARING:
Plan to Share IPD: No
Basic, de-identified individual participant data will be made available once all data collection and analysis is complete